CLINICAL TRIAL: NCT03248778
Title: Readiness to Disclose Mother's HIV Diagnosis to Their Children in Beijing, China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000020567
Record Dates: First submitted 2017-08-10; First posted 2017-08-14 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: HIV
Keywords: disclosure

STUDY DESIGN:
Intervention Model Description: The investigators will assess feasibility and acceptability and get a broad sense of the initial efficacy of the intervention with a two-arm RCT implemented with 10 HIV+ mothers: 5 will be randomly assigned to the disclosure-support counseling intervention and 5 to a treatment-as-usual (TAU) condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- disclosure-support counseling (Experimental)
  Interventions: Behavioral: disclosure-support counseling intervention
- Treatment as Usual (No Intervention)

INTERVENTIONS:
Behavioral: disclosure-support counseling intervention — The intervention will include three components: (a) assessment; (b) decision-making and support; and (c) disclosure, planning, and action. The individualized assessment comprehensively will consider the family's history, experiences with disclosure, communication skills, coping resources, and factors likely to affect disclosure (e.g., familial, psychological, social, cultural, and medical issues). The second component of decision-making and support focused on developing communication skills and strategies, with role-play and practice outside of the sessions as necessary. Costs and benefits of disclosure were considered along with the range of disclosure options. Materials, including a pros and cons chart of disclosure and a disclosure continuum worksheet, were used to stimulate discussions of possible plans and consequences. In the third component, parents were encouraged to formulate and practice a disclosure plan for later use.
  Arms: disclosure-support counseling

SUMMARY:
Specific aims of the 1-year project are to pilot test the disclosure support intervention by (a) evaluating acceptability and feasibility with a preliminary randomized trial among 10 HIV+ mothers (5 in the intervention group and 5 in the treatment as usual (TAU) group) and (b) assessing outcomes in mothers (quality of life and mental health indicators, adherence, social support, and disclosure stress, efficacy, readiness, and completion). The intervention will be compared to treatment as usual, with baseline (0 weeks), immediate post-intervention (4 weeks), and 12-week follow-up (16 weeks) assessments.

DETAILED DESCRIPTION:
HIV disclosure to children has been shown to strengthen family relations and increase assistance with medical care, reinforcing the parent's willingness to live. Some Chinese children aware of their parents HIV diagnosis do exhibit emotional and social dysfunction; however, adequate support from caregivers (e.g., grandparents or even their HIV+ parents) can improve the children's quality of life and academic performance. There is a clear need for practical interventions to address parental distress around HIV disclosure in China, where cultural norms often emphasize family identity and cohesion and underscore the need for family-based programs, which have been shown to be feasible and efficacious for HIV-affected families.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ mother ≥18 years of age,
* not psychotic or demented;
* receiving clinical care at the Ditan hospital,
* a mother of an HIV-negative child of age 13-25 years who does not know about the mother's infection;
* well enough to attend study sessions as the clinic.

Exclusion Criteria:

* no psychotic or demented

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
readiness to disclose | 16 weeks
  This data will be collected and evaluated with qualitative methods using the Disclosure Distress Questionnaire

SECONDARY OUTCOMES:
quality of life via Medical Outcomes Study HIV Health Survey | 16 weeks
  The Medical Outcomes Study HIV Health Survey (MOS-HIV) is a brief, comprehensive health status measure that has been used extensively in studies of human immunodeficiency virus/acquired immune deficiency syndrome (HIV/AIDS). MOS-HIV for quality of life is ranges from 0-60. The higher the score the better the quality of life.
depression via the Center for Epidemiologic Studies Depression Scale (CES-D) | 16 weeks
  Depression is measured by CES-D, ranged from 0-40. A score higher than 16 is considered as depressed.
adherence | 16 weeks
  Measured using a visual analog scale. Acceptable adherence is equal or higher than 95%.
social support using the HIV Social Support tool | 16 weeks
  social support will ranged from 0-20. The higher the score, shown more support in life.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Ti Chen, PhD, Principal Investigator — Yale School of Nursing
Locations (1):
- Beijing Ditan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No